CLINICAL TRIAL: NCT05169424
Title: Comparison of Exacerbation Risk and Health Outcomes in Maintenance Treatment naïve Chronic Obstructive Pulmonary Disease (COPD) Patients Using Stiolto Versus Trelegy, a Real-World Study
Brief Title: A Study in the US Based on Pharmacy and Medical Claims That Compares How Well Stiolto® and Trelegy® Work in People With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0121
Record Dates: First submitted 2021-12-02; First posted 2021-12-27 (Actual); Results first posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2022-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol; fluticasone furoate; GSK573719; vilanterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Stiolto initiators: Chronic obstructive pulmonary disease (COPD) patients who initiated with Stiolto Respimat (Tiotropium + Olodaterol (5/5 micrograms (mcg)) in the existing real-world data from the Commercial Insurance and Medicare beneficiaries data using administrative claims between 15 September 2016 and 31st March 2020.
  All participants had enrolled 1 year before the index date (starting from 15 September 2017).
  Interventions: Device: Stiolto Respimat; Drug: Tiotropium + Olodaterol (5/5 mcg)
- Trelegy initiators: COPD patients who initiated with Trelegy Ellipta (Fluticasone Furoate + Umeclidinium + Vilanterol (100/62.5/25 mcg) in the existing real-world data from the Commercial Insurance and Medicare beneficiaries data using administrative claims between 15 September 2016 and 31st March 2020.
  All participants had enrolled 1 year before the index date (starting from 15 September 2017).
  Interventions: Device: Trelegy Ellipta; Drug: Fluticasone Furoate + Umeclidinium + Vilanterol (100/62.5/25 mcg)

INTERVENTIONS:
Device: Trelegy Ellipta — Trelegy Ellipta
  Groups: Trelegy initiators
Device: Stiolto Respimat — Stiolto Respimat
  Groups: Stiolto initiators
Drug: Tiotropium + Olodaterol (5/5 mcg) — Tiotropium + Olodaterol (5/5 mcg)
  Groups: Stiolto initiators
Drug: Fluticasone Furoate + Umeclidinium + Vilanterol (100/62.5/25 mcg) — Fluticasone Furoate + Umeclidinium + Vilanterol (100/62.5/25 mcg)
  Groups: Trelegy initiators

SUMMARY:
This study looks at data from people with chronic obstructive pulmonary disease (COPD). Some used Stiolto Respimat and the others Trelegy Ellipta as their first treatment for COPD.

The purpose of this study is to find out how well the treatments worked. Researchers compare the time to first COPD flare-up (exacerbation) between the 2 treatments.

The study analyses anonymous data from pharmacy claims collected over 3.5 years.

ELIGIBILITY:
Inclusion Criteria:

* ≥40 years of age as of the year of the index date
* At least one pharmacy claim for Stiolto Respimat or Trelegy Ellipta.

  * For Stiolto Respimat users, the first pharmacy claim of Fixed Dose Combination (FDC) of Tiotropium + Olodaterol (5/5 micrograms (mcg)) will be defined as the index date.
  * For Trelegy Ellipta users, the first pharmacy claim of FDC of Fluticasone Furoate + Umeclidinium + Vilanterol (100/62.5/25 mcg), will be defined as the index date.
* Two medical claims (at least one claim on index date or before in the baseline period) with an International Statistical Classification of Diseases and Related Health Problems (ICD)-9/10 diagnosis code(s) for chronic obstructive pulmonary disease (COPD) in any position during the study period (baseline ± post index date).
* At least one year of continuous medical and pharmacy health plan eligibility prior to the index date is required (to allow a baseline period for the covariates and characterizing the study population).

Exclusion Criteria:

* To increase the likelihood of a true diagnosis of COPD, we will exclude all patients with two medical claims of asthma, cystic fibrosis, lung cancer, or interstitial lung disease in any position on separate dates of service during the study period.
* To restrict the cohort to first line maintenance therapy of Stiolto Respimat or first line maintenance therapy of Trelegy Ellipta we will exclude: patients on long-acting muscarinic antagonists (LAMA) monotherapy; long-acting beta2 agonists (LABA) monotherapy; inhaled corticosteroids (ICS) monotherapy; free or FDC of: ICS+LABA, LAMA+LABA, ICS+LABA+LAMA therapy within six months prior to index date.
* Pharmacy claims for multiple index medications on the index date.
* Pharmacy claims for non-index COPD maintenance medications on the index date.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample will include medical and pharmacy claim records for COPD patients included in the IQVIA database (previously named IMS Pharmetrix).
Sampling Method: Non-Probability Sample
Enrollment: 9117 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2021-12-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- eMax health, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- [Derived] Shaikh A, Ritz J, Casciano J, Palli SR, Clark B, Dotiwala Z, Quint JK. Clinical and Economic Evaluation of Fluticasone Furoate/Umeclidinium/Vilanterol Versus Tiotropium/Olodaterol Therapy in Maintenance Treatment-Naive Patients with COPD in the US. Int J Chron Obstruct Pulmon Dis. 2025 Feb 14;20:335-348. doi: 10.2147/COPD.S479504. eCollection 2025. PMID 39968202
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional, observational, retrospective study using existing real-world data, investigating the risk of Chronic obstructive pulmonary disease (COPD) exacerbations, community acquired pneumonia, and health care utilization in maintenance treatment naive patients treated as first line therapy with Stiolto, in comparison to Trelegy.
Pre-assignment Details: All subjects who strictly met all inclusion and none of the exclusion criteria were included.
Period: Overall Study
Arm/Group | Stiolto Initiators | Trelegy Initiators
Started | 3996 | 5121
Propensity Score Matching | 2951 | 2951
Completed | 3996 | 5121
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who strictly met all inclusion and none of the exclusion criteria were included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stiolto Initiators | Trelegy Initiators | Total
Number analyzed (Participants) | 3996 | 5121 | 9117
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (8.37) | 60.9 (78.7) | 61.25 (8.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1894 | 2368 | 4262
  Male | 2102 | 2753 | 4855
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Chronic Obstructive Pulmonary Disease (COPD) Exacerbation After Cohort Entry
Description: Incidence rate of chronic obstructive pulmonary disease (COPD) exacerbation after cohort entry were reported. The incidence rate was calculated as totaling the number of exacerbation for all patients / total follow-up in days * 365.
Time Frame: From index date (i.e. baseline, cohort entry, 15 September 2017) until 31st March 2020, up to 30 months and 16 days.
Population: Only subjects who strictly met all inclusion and none of the exclusion criteria and who were included in the propensity score matched cohort.
Measure: Number; unit: exacerbation per patient-year
Arm/Group | Stiolto Initiators | Trelegy Initiators
Number analyzed (Participants) | 2951 | 2951
exacerbation per patient-year | 0.28 | 0.32
Statistical Analysis 1: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other — Comparison of Stiolto (reference group) versus Trelegy for incidence rate of exacerbation; p = 0.064, Regression, Cox; Cox regression was for time to first exacerbation and cohort as covariate; Hazard Ratio (HR) = 1.133, 95% CI 2-sided [0.993 to 1.293]
Statistical Analysis 2: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other; p = 0.045, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other; p = 0.063, Log Rank

2. Primary Outcome: Incidence Rate of Chronic Obstructive Pulmonary Disease (COPD) Exacerbation After Cohort Entry - Among Patients With no Baseline Exacerbation
Description: Incidence rate of chronic obstructive pulmonary disease (COPD) exacerbation after cohort entry among patients with no baseline exacerbation were reported. The incidence rate was calculated as totaling the number of exacerbation for all patients / total follow-up in days * 365.
Time Frame: From index date (i.e. baseline, cohort entry, 15 September 2017) until 31st March 2020, up to 30 months and 16 days.
Population: Only subjects who strictly met all inclusion and none of the exclusion criteria and who were included in the propensity score matched cohort. Only subject who had no baseline exacerbation were included in the analysis.
Measure: Number; unit: exacerbation per patient-year
Arm/Group | Stiolto Initiators | Trelegy Initiators
Number analyzed (Participants) | 2128 | 2114
exacerbation per patient-year | 0.25 | 0.3
Statistical Analysis 1: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other — Comparison of Stiolto (reference group) versus Trelegy; p = 0.057, Regression, Cox; Cox regression was for time to first exacerbation and cohort as covariate; Hazard Ratio (HR) = 1.169, 95% CI 2-sided [0.996 to 1.372]

3. Primary Outcome: Incidence Rate of Chronic Obstructive Pulmonary Disease (COPD) Exacerbation After Cohort Entry - Among Patients With 0 or 1 Baseline Exacerbation
Description: Incidence rate of chronic obstructive pulmonary disease (COPD) exacerbation after cohort entry among patients with 0 or 1 baseline exacerbation were reported. The incidence rate was calculated as totaling the number of exacerbation for all patients / total follow-up in days * 365.
Time Frame: From index date (i.e. baseline, cohort entry, 15 September 2017) until 31st March 2020, up to 30 months and 16 days.
Population: Only subjects who strictly met all inclusion and none of the exclusion criteria and who were included in the propensity score matched cohort. Only subject who had 0 or 1 baseline exacerbation were included in the analysis.
Measure: Number; unit: exacerbation per patient-year
Arm/Group | Stiolto Initiators | Trelegy Initiators
Number analyzed (Participants) | 2852 | 2829
exacerbation per patient-year | 0.27 | 0.31
Statistical Analysis 1: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other — Comparison of Stiolto (reference group) versus Trelegy; p = 0.114, Regression, Cox; Cox regression was for time to first exacerbation and cohort as covariate; Hazard Ratio (HR) = 1.116, 95% CI 2-sided [0.974 to 1.279]

4. Primary Outcome: Incidence Rate of Chronic Obstructive Pulmonary Disease (COPD) Exacerbation After Cohort Entry - Among Patients With 2 or More Baseline Exacerbations
Description: Incidence rate of chronic obstructive pulmonary disease (COPD) exacerbation after cohort entry among patients with 2 or more baseline exacerbations were reported. The incidence rate was calculated as totaling the number of exacerbation for all patients / total follow-up in days * 365.
Time Frame: From index date (i.e. baseline, cohort entry, 15 September 2017) until 31st March 2020, up to 30 months and 16 days.
Population: Only subjects who strictly met all inclusion and none of the exclusion criteria and who were included in the propensity score matched cohort. Only subjects with 2 or more baseline exacerbations were included in the analysis.
Measure: Number; unit: exacerbation per patient-year
Arm/Group | Stiolto Initiators | Trelegy Initiators
Number analyzed (Participants) | 99 | 122
exacerbation per patient-year | 0.49 | 0.58
Statistical Analysis 1: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other — Comparison of Stiolto (reference group) versus Trelegy; p = 0.273, Regression, Cox; Cox regression was for time to first exacerbation and cohort as covariate; Hazard Ratio (HR) = 1.374, 95% CI 2-sided [0.779 to 2.424]

5. Secondary Outcome: Incidence Rate of Pneumonia Hospitalization (Diagnosis in Any Position)
Description: The incidence rates of pneumonia (pneu.) hospitalization (diagnosis in any position) were reported. The incidence rate was calculated as totaling the number of pneumonia hospitalization for all patients / total follow-up in days * 365.
Time Frame: From index date (i.e. baseline, cohort entry, 15 September 2017) until 31st March 2020, up to 30 months and 16 days.
Population: as for outcome 1
Measure: Number; unit: pneu. hospitalization per patient-year
Arm/Group | Stiolto Initiators | Trelegy Initiators
Number analyzed (Participants) | 2951 | 2951
pneu. hospitalization per patient-year | 0.025 | 0.030
Statistical Analysis 1: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other — Comparison of Stiolto (reference) versus Trelegy for incidence rate of pneumonia hospitalization; p = 0.429, Regression, Cox; Hazard Ratio (HR) = 1.183, 95% CI 2-sided [0.780 to 1.792]
Statistical Analysis 2: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other; p = 0.896, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other; p = 0.932, Log Rank

6. Secondary Outcome: Incidence Rate of Pneumonia Hospitalization (Diagnosis in Any Position) - Among Patients With no Baseline Exacerbation
Description: The incidence rates of pneumonia (pneu.) hospitalization (diagnosis in any position) among patients with no baseline exacerbation were reported. The incidence rate was calculated as totaling the number of pneumonia hospitalization for all patients / total follow-up in days * 365.
Time Frame: From index date (i.e. baseline, cohort entry, 15 September 2017) until 31st March 2020, up to 30 months and 16 days.
Population: Only subjects who strictly met all inclusion and none of the exclusion criteria and who were included in the propensity score matched cohort. Only participants with no baseline exacerbation were included.
Measure: Number; unit: pneu. hospitalization per patient-year
Arm/Group | Stiolto Initiators | Trelegy Initiators
Number analyzed (Participants) | 2128 | 2114
pneu. hospitalization per patient-year | 0.024 | 0.023
Statistical Analysis 1: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other — Comparison of Stiolto (reference) versus Trelegy for incidence rate of pneumonia hospitalization; p = 0.935, Regression, Cox; Hazard Ratio (HR) = 0.979, 95% CI 2-sided [0.582 to 1.645]

7. Secondary Outcome: Incidence Rate of Pneumonia Hospitalization (Diagnosis in Any Position) - Among Patients With 0 or 1 Baseline Exacerbation
Description: The incidence rates of pneumonia (pneu.) hospitalization (diagnosis in any position) among patients with 0 or 1 baseline exacerbation were reported. The incidence rate was calculated as totaling the number of pneumonia hospitalization for all patients / total follow-up in days * 365.
Time Frame: From index date (i.e. baseline, cohort entry, 15 September 2017) until 31st March 2020, up to 30 months and 16 days.
Population: Only subjects who strictly met all inclusion and none of the exclusion criteria and who were included in the propensity score matched cohort. Only participants with 0 or 1 baseline exacerbation were included.
Measure: Number; unit: pneu. hospitalization per patient-year
Arm/Group | Stiolto Initiators | Trelegy Initiators
Number analyzed (Participants) | 2852 | 2829
pneu. hospitalization per patient-year | 0.024 | 0.028
Statistical Analysis 1: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other — Comparison of Stiolto (reference) versus Trelegy for incidence rate of pneumonia hospitalization; p = 0.507, Regression, Cox; Hazard Ratio (HR) = 1.159, 95% CI 2-sided [0.750 to 1.790]

8. Secondary Outcome: Incidence Rate of Pneumonia Hospitalization (Diagnosis in Any Position) - Among Patients With 2 or More Baseline Exacerbations
Description: The incidence rates of pneumonia (pneu.) hospitalization (diagnosis in any position) among patients with 2 or more baseline exacerbations were reported. The incidence rate was calculated as totaling the number of pneumonia hospitalization for all patients / total follow-up in days * 365.
Time Frame: From index date (i.e. baseline, cohort entry, 15 September 2017) until 31st March 2020, up to 30 months and 16 days.
Population: Only subjects who strictly met all inclusion and none of the exclusion criteria and who were included in the propensity score matched cohort. Only participants with 2 or more baseline exacerbations were included.
Measure: Number; unit: pneu. hospitalization per patient-year
Arm/Group | Stiolto Initiators | Trelegy Initiators
Number analyzed (Participants) | 99 | 122
pneu. hospitalization per patient-year | 0.075 | 0.072
Statistical Analysis 1: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other — Comparison of Stiolto (reference) versus Trelegy for incidence rate of pneumonia hospitalization; p = 0.726, Regression, Cox; Hazard Ratio (HR) = 1.291, 95% CI 2-sided [0.309 to 5.405]

9. Secondary Outcome: Total Costs of COPD or Pneumonia-related Health Care Cost and Resource Utilization (HCRU)
Description: The total annualized costs of COPD or pneumonia-related health care cost and resource utilization (HCRU) were calculated for each cohort by totaling the costs for all patients divided by the total follow-up in days, multiplied by 365.
Time Frame: From index date (i.e. baseline, cohort entry, 15 September 2017) until 31st March 2020, up to 30 months and 16 days.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: dollars per year
Arm/Group | Stiolto Initiators | Trelegy Initiators
Number analyzed (Participants) | 2951 | 2951
dollars per year | 9834 [8413 to 11256] | 10020 [8216 to 11824]
Statistical Analysis 1: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other; p = 0.874, t-test, 2 sided
Statistical Analysis 2: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other; p = 0.01, ZINB regression with log link; The costs were modeled using Zero Inflated Negative Binomial (ZINB) regression with log link with cohort as the only covariate; Exponential estimate = 0.895, 95% CI 2-sided [0.823 to 0.974] — The analysis was for Stiolto versus Trlegy (Trelegy was the reference group)

10. Secondary Outcome: Total Costs of COPD-related HCRU
Description: The total annualized costs of COPD-related HCRU were calculated for each cohort by totaling the costs for all patients divided by the total follow-up in days, multiplied by 365.
Time Frame: From index date (i.e. baseline, cohort entry, 15 September 2017) until 31st March 2020, up to 30 months and 16 days.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: dollars per year
Arm/Group | Stiolto Initiators | Trelegy Initiators
Number analyzed (Participants) | 2951 | 2951
dollars per year | 9688 [8271 to 11105] | 9834 [8038 to 11630]
Statistical Analysis 1: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other; p = 0.899, t-test, 2 sided
Statistical Analysis 2: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other; p = 0.012, ZINB regression with log link; [statistical method as in outcome 9, analysis 2]; Exponential estimate = 0.897, 95% CI 2-sided [0.824 to 0.976] — The analysis was for Stiolto versus Trlegy (Trelegy was the reference group)

11. Secondary Outcome: Total Costs of Pneumonia-related HCRU
Description: The total annualized costs of pneumonia-related HCRU were calculated for each cohort by totaling the costs for all patients divided by the total follow-up in days, multiplied by 365.
Time Frame: From index date (i.e. baseline, cohort entry, 15 September 2017) until 31st March 2020, up to 30 months and 16 days.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: dollars per year
Groups:
- Stiolto Initiators: Chronic obstructive pulmonary disease (COPD) patients who initiated with Stiolto Respimat (Tiotropium + Olodaterol (5/5 micrograms (mcg)) in the existing real-world data from the Commercial Insurance and Medicare beneficiaries data using administrative claims between 15 September 2016 and 31st March 2020.
- Trelegy Initiators: COPD patients who initiated with Trelegy Ellipta (Fluticasone Furoate + Umeclidinium + Vilanterol (100/62.5/25 mcg) in the existing real-world data from the Commercial Insurance and Medicare beneficiaries data using administrative claims between 15 September 2016 and 31st March 2020.
Arm/Group | Stiolto Initiators | Trelegy Initiators
Number analyzed (Participants) | 2951 | 2951
dollars per year | 2244 [1406 to 3082] | 2274 [676 to 3872]
Statistical Analysis 1: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other; p = 0.974, t-test, 2 sided
Statistical Analysis 2: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other; p = 0.595, ZINB regression with log link; [statistical method as in outcome 9, analysis 2]; Exponential estimate = 1.135, 95% CI 2-sided [0.711 to 1.812] — The analysis was for Stiolto versus Trlegy (Trelegy was the reference group)

12. Secondary Outcome: Total Costs of COPD or Pneumonia Attributable HCRU
Description: The total annualized costs of COPD or pneumonia attributable HCRU were calculated for each cohort by totaling the costs for all patients divided by the total follow-up in days, multiplied by 365.
Time Frame: From index date (i.e. baseline, cohort entry, 15 September 2017) until 31st March 2020, up to 30 months and 16 days.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: dollars per year
Arm/Group | Stiolto Initiators | Trelegy Initiators
Number analyzed (Participants) | 2951 | 2951
dollars per year | 5729 [4565 to 6894] | 5409 [4808 to 6009]
Statistical Analysis 1: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other; p = 0.622, t-test, 2 sided
Statistical Analysis 2: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other; p = 0.855, ZINB regression with log link; [statistical method as in outcome 9, analysis 2]; Exponential estimate = 1.008, 95% CI 2-sided [0.928 to 1.094] — The analysis was for Stiolto versus Trlegy (Trelegy was the reference group)

13. Secondary Outcome: Total Costs of All-cause HCRU
Description: The total annualized costs of all-cause HCRU were calculated for each cohort by totaling the costs for all patients divided by the total follow-up in days, multiplied by 365.
Time Frame: From index date (i.e. baseline, cohort entry, 15 September 2017) until 31st March 2020, up to 30 months and 16 days.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: dollars per year
Arm/Group | Stiolto Initiators | Trelegy Initiators
Number analyzed (Participants) | 2951 | 2951
dollars per year | 20849 [18803 to 22896] | 19384 [17282 to 21487]
Statistical Analysis 1: Comparison: Stiolto Initiators vs Trelegy Initiators; Test type: Other; p = 0.328, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study
Description: As this is a non-interventional study with secondary use of existing real-world data from the Commercial Insurance and Medicare beneficiaries data using administrative claims, safety monitoring and safety reporting on an individual case level is not applicable. The "0" in All-cause Mortality, Serious Adverse Events, and Other Adverse Events sections indicates "not applicable".
Arm/Group | Stiolto Initiators | Trelegy Initiators
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT05169424/Prot_SAP_000.pdf